CLINICAL TRIAL: NCT05190328
Title: Effects Of Muscle Energy Technique Versus Active Release Technique On Pain, Cervical Range Of Motion And Functional Disability In Patients With Upper Cross Syndrome: A Randomized Controlled Trial.
Brief Title: Muscle Energy Technique Versus Active Release Technique on Pain, Cervical Range Of Motion And Functional Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Anam Akram, EFFECTS OF MUSCLE ENERGY TECHNIQUE VERSUS ACTIVE RELEASE TECHNIQUE ON PAIN, CERVICAL RANGE OF MOTION AND FUNCTIONAL DISABILITY IN PATIENTS WITH UPPER CROSS SYNDROME: A RANDOMIZED CONTROLLED TRIAL., University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/980/2021
Record Dates: First submitted 2021-12-30; First posted 2022-01-13 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Upper Cross Syndrome
Keywords: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (Experimental): Experimental: Muscle Energy Technique Post isometric relaxation: Patient will perform isometrics on upper trapezius and levator scapulae one by one. Each isometric contraction will be held for 10 seconds and then participants will be asked to relax the contraction with exhalation. This will be repeated five times in one session.
  Routine Physical Therapy including TENS, Hot Pack, Strengthening, and stretching exercises will also be delivered along with the Muscle energy technique.
  Interventions: Other: Muscle Energy Technique
- Active Release Technique (Experimental): Experimental: Active Release Technique: The therapist will apply deep pressure on both sides of levator scapulae and upper trapezius muscles (over the area of tenderness) and the patient will be instructed to actively move the muscle from a shortened to lengthened position and thereby breaking adhesions.1 set of 5 repetitions in one session.
  Routine Physical Therapy including TENS, Hot Pack, Strengthening, and stretching exercises will also be delivered along with active release technique
  Interventions: Other: Active Release Technique

INTERVENTIONS:
Other: Muscle Energy Technique — Experimental: Muscle Energy Technique Post isometric relaxation: Patient will perform isometrics on upper trapezius and levator scapulae one by one. Each isometric contraction will be held for 10 seconds and then participants will be asked to relax the contraction with exhalation. This will be repeated five times in one session.
  Routine Physical Therapy including TENS, Hot Pack, Strengthening, and stretching exercises will also be delivered along with Muscle energy technique.
  Arms: Muscle Energy Technique
Other: Active Release Technique — Experimental: Active Release Technique: Therapist will apply deep pressure on both sides of levator scapulae and upper trapezius muscles (over the area of tenderness) and the patient is instructed to actively move the muscle from the shortened to a lengthened position and thereby breaking adhesions. 1 set of 5 repetitions in one session.
  Routine Physical Therapy including TENS, Hot Pack, Strengthening, and stretching exercises will also be delivered along with Active Release Technique.
  Arms: Active Release Technique

SUMMARY:
The study will be a randomized controlled trial. This study will be conducted in The University of Lahore Teaching Hospital, Lahore, Pakistan. A sample size of 86 will be randomly allocated into two experimental groups,(43 participants in each group), by using computer-generated random number list method. The participants randomly allocated into two experimental, group A will receive Muscle energy technique (METs) specifically, Post isometric relaxation technique for upper trapezius and levator scapulae muscles, 1 set of 5 repetitions and 10 seconds hold along with routine physical therapy as (Hot pack, transcutaneous electrical nerve stimulator, strengthening and stretching exercises).

Experimental group B will be delivered Active Release Technique on both sides of levator scapulae and upper trapezius muscles 1 set of 5 repetitions along with routine physical therapy as (Hot pack, transcutaneous electrical nerve stimulator, strengthening and stretching exercises).

Both experimental groups will receive twelve treatment sessions (3 sessions per week for 4 weeks)

DETAILED DESCRIPTION:
Recruitment: Participants will be recruited and referred by orthopedic doctor from The University of Lahore Teaching Hospital to Physical Therapy Department.

Randomization and Allocation: The participants after confirming the eligibility criteria will be randomly allocated into two experimental groups (Group A, Group B) by using computer generated random number list method.

Blindness: The study will be single blinded, and an independent investigator will perform randomization and will inform the patients and the therapist about the allocation of participants and assessor will be blinded.

Intervention: The participants will be randomly allocated into two experimental groups (Group A, Group B). Experimental Group A will receive Muscle energy technique (METs) specifically, Post isometric relaxation technique for upper trapezius and levator scapulae muscles, 1 set of 5 repetitions, and 10 seconds hold along with routine physical therapy as (Hot pack, transcutaneous electrical nerve stimulator, strengthening and stretching exercises).

Experimental group B will be delivered Active Release Technique on both sides of levator scapulae and upper trapezius muscles 1 set of 5 repetitions along with routine physical therapy as (Hot pack, TENS, strengthening and stretching exercises).

Duration:Both experimental groups will receive twelve treatment sessions (3 sessions per week for 4 weeks, each session of 35-45 minutes)

Outcome Variables and Measures:

Pain (Numeric Pain Rating Scale) Range of Motion (Universal Goniometer) Functional Disability (Neck disability Index Questionnaire) Outcome measures will be taken at baseline, end of 6th treatment session (2nd week), end of 12th session (4th week) and follow up will be obtained after 1 month (8th week) and then collected data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • The diagnosed Upper cross syndrome patients aged 20-35 years will be included in this study

  * Both male and females will be included in this study.
  * Patients with pain of at least 3 points on NPRS.
  * The participants with neck disability of at least 10/50 on the Neck Disability Index (NDI) will be included in this study.

Exclusion Criteria:

* • Cervical radiculopathy or myelopathy.

  * History of trauma, whiplash injury, cervical instability or fractures in cervical spine.
  * Systemic illness i.e. cardiovascular disorders, respiratory disorders etc.
  * Inflammatory disease i.e. rheumatoid arthritis, ankylosing spondylitis, osteomyelitis.
  * Any pathology i.e. infection, osteoporosis, malignancy bony disease i.e. osteosarcoma.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  The Numeric pain rating scale (NPRS) is self-reported and simple tool to measure level of pain. This is 11-point numeric scale in this scale the respondents will select the intensity of their pain ranging from 0-10, where 0 means no pain and 10 means severe pain
Neck Disability Index (NDI) questionnaire | 4 weeks
  The neck disability index (NDI) questionnaire is comprise of 10 items and is frequently used as a patient reported outcome measurement tool to evaluate the physical and functional capacity of an individual with cervical pain.Neck disability index is also used to evaluate the difference between pre and post treatment. Each section on NDI is scored on 0 to 5 rating in which 0 points or 0% means no pain or no activity limitation and 5 means worst imaginable pain or 50 points or 100% means complete activity limitation.
Range of motion | 4 weeks
  Universal Goniometer is a clinical and easily available tool which is commonly used by physiotherapist to document the available range of movement at certain joints.

CONTACTS AND LOCATIONS:
Overall Officials: Anam Akram, MS-MSK*, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karimian R, Rahnama N, Ghasemi G, Lenjannejadian S. Photogrammetric Analysis of Upper Cross Syndrome among Teachers and the Effects of National Academy of Sports Medicine Exercises with Ergonomic Intervention on the Syndrome. J Res Health Sci. 2019 Jul 3;19(3):e00450. PMID 31586371
- [Background] Kang JI, Choi HH, Jeong DK, Choi H, Moon YJ, Park JS. Effect of scapular stabilization exercise on neck alignment and muscle activity in patients with forward head posture. J Phys Ther Sci. 2018 Jun;30(6):804-808. doi: 10.1589/jpts.30.804. Epub 2018 Jun 12. PMID 29950768
- [Background] Kim JH, Lee HS, Park SW. Effects of the active release technique on pain and range of motion of patients with chronic neck pain. J Phys Ther Sci. 2015 Aug;27(8):2461-4. doi: 10.1589/jpts.27.2461. Epub 2015 Aug 21. PMID 26357426
- [Background] Thomas E, Cavallaro AR, Mani D, Bianco A, Palma A. The efficacy of muscle energy techniques in symptomatic and asymptomatic subjects: a systematic review. Chiropr Man Therap. 2019 Aug 27;27:35. doi: 10.1186/s12998-019-0258-7. eCollection 2019. PMID 31462989
- [Background] Gillani SN, Ain Q-, Rehman SU, Masood T. Effects of eccentric muscle energy technique versus static stretching exercises in the management of cervical dysfunction in upper cross syndrome: a randomized control trial. J Pak Med Assoc. 2020 Mar;70(3):394-398. doi: 10.5455/JPMA.300417. PMID 32207413